CLINICAL TRIAL: NCT06860607
Title: Environment and Alcohol: A Pilot Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10002341; 002341-DA
Record Dates: First submitted 2025-03-05; First posted 2025-03-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-21

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Economics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject with alcohol use disorder (Other): subjects (Female/ Male) aged 21 and up
  Interventions: Behavioral: Evaluate the effects of Environmental Enrichment (EE) on alcohol consumption

INTERVENTIONS:
Behavioral: Evaluate the effects of Environmental Enrichment (EE) on alcohol consumption — This study investigates how different environments and activities affect alcohol consumption and related outcomes.

SUMMARY:
Background:

Alcohol use disorder (AUD) is a chronic disease that causes more than 140,000 US deaths each year. AUD treatment often includes therapy and medication. Some people with AUD may also benefit from behavioral and lifestyle changes.

Objective:

To evaluate the effects of different activities and environments on drinking behaviors and mental health in people with AUD.

Eligibility:

People aged 21 years and older with AUD.

Design:

Participants will have up to 10 study visits in Baltimore.

Participants will have a baseline visit. They will have a physical exam with blood and urine tests. They will have a breath test for alcohol and a test that measures body composition. They will answer questions about their alcohol and substance use; mental and physical health; mood and anxiety; and sleep quality.

Participants will download an app called MetricWire. The app will send 3 sets of questions to be answered at different times throughout the day.

The study visits will include 2 stages:

1. Active stage. On these visits, participants will use a virtual reality system called the Meta Quest Pro (MQP) as they choose. Then they may choose among video games, puzzles, books, crafts, and other activities.. These sessions will last for 3 hours.
2. Passive stage. On these visits, participants will watch videos selected by the research team. These sessions will last for 3 hours.

On the last visit of each stage, participants will sit in a room that looks like a bar. They will answer questions about their cravings, their urge to drink, and how many drinks they would buy. Participants will be served 1 drink containing alcohol. They will be asked about their cravings and subjective effects of alcohol after drinking it.

DETAILED DESCRIPTION:
Study Description:

This study will investigate the effects of cognitive and sensorimotor environmental enrichment (EE) on alcohol drinking, alcohol cue-reactivity, and other related outcomes in participants with alcohol use disorder (AUD). The hypothesis is that the psychological and physiological effects of environmental enrichment will confer therapeutic benefits for people with AUD, especially on measures of alcohol consumption and cue-elicited craving.

Objectives:

Primary Objectives:

1. Evaluate the effects of EE on alcohol consumption

Secondary Objectives:

1. Evaluate the effects of EE on other ecological momentary assessments (EMA)
2. Evaluate the effects of EE on bar-lab assessments

Endpoints:

Primary Endpoints:

1. Self-reported alcohol consumed using ecological momentary assessment

Secondary Endpoints:

1. State assessments of varying psychological, social, and environmental domains associated with AUD
2. - Cue reactivity: AUQ, AAS

   * APT
   * Alcohol challenge: B-BAES, DEQ-5, AUQ, BrAC

ELIGIBILITY:
* INCLUSION CRITERIA:

To meet eligibility for this study, participants must meet all the following criteria:

1. At least 21 years old
2. Owns a cellular device ("smart phone") and is willing to download the EMA application and use it to answer the study questionnaires
3. Diagnosis of alcohol use disorder (minimum of 2 DSM-5 criteria on a valid diagnostic tool, e.g., Mini-International Neuropsychiatric Interview (MINI) or the Structured Clinical Interview for DSM Disorders (SCID))
4. Self-reported drinking, according to alcohol Timeline Follow-Back (TLFB), of > 7 drinks per week for females or > 14 drinks per week for males, on average, during the 28-day period prior to screening + at least four days with > 3 drinks for females or > 4 drinks for males during the 28-day period prior to screening
5. Most recent Clinical Institute Withdrawal Assessment for Alcohol - revised (CIWA-Ar) score < 10
6. If a female of childbearing potential: not pregnant or breastfeeding, no intention to become pregnant during the study duration, and agrees to use a highly effective contraception method to prevent pregnancy for the entire study duration. Highly effective contraception methods will be determined by the MAI or designee.

EXCLUSION CRITERIA:

Any individual who meets any of the following criteria will be excluded from this study:

1. Current use of FDA-approved pharmacotherapy for AUD (or of a medication intended as an off-label use to treat AUD as determined by the MAI), or currently seeking treatment for AUD
2. Medical and/or mental health conditions that are clinically unstable and would therefore compromise the safety and/or scientific integrity of the study, as determined by the MAI or study team respectively.
3. Known history of clinically significant cybersickness.
4. Any other reason or clinical condition that the Investigators judge would interfere with study participation and/or be unsafe for a participant
5. Unable to speak, read, write, and understand English

Justification: Many of the assessments have only been validated in English, and therefore, a non-English translation would jeopardize the scientific integrity of the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effects of EE on alcohol consumption | 1-3 months for each participant
  Self-reported alcohol consumed using ecological momentary assessment

SECONDARY OUTCOMES:
Evaluate the effects of EE on other EMA assessments | 1-3 months for each participant
  Real-time, real-world data collection of state variables and alcohol consumption enhances the ecological validity of the data. This also allows for evaluation of how dynamics in psychological, social and environmental measures are related to changes in alcohol consumption.
Evaluate the effects of EE on bar-lab assessments | 1-3 months for each participant
  Alcohol craving (measure here via AUQ) is a key factor and predictor of persistent and heavy alcohol use and is attenuated by some treatments. AAS measures attention to alcohol cues. APT serves as a measure of economic demand for alcohol. The subjective response to alcohol is a predictor of AUD vulnerability and treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koob GF, Volkow ND. Neurobiology of addiction: a neurocircuitry analysis. Lancet Psychiatry. 2016 Aug;3(8):760-773. doi: 10.1016/S2215-0366(16)00104-8. PMID 27475769
- [Background] Nicastri CM, McFeeley BM, Simon SS, Ledreux A, Hakansson K, Granholm AC, Mohammed AH, Daffner KR. BDNF mediates improvement in cognitive performance after computerized cognitive training in healthy older adults. Alzheimers Dement (N Y). 2022 Aug 30;8(1):e12337. doi: 10.1002/trc2.12337. eCollection 2022. PMID 36089933
- [Background] Nithianantharajah J, Hannan AJ. Enriched environments, experience-dependent plasticity and disorders of the nervous system. Nat Rev Neurosci. 2006 Sep;7(9):697-709. doi: 10.1038/nrn1970. PMID 16924259
- [Background] Edwards S, Kenna GA, Swift RM, Leggio L. Current and promising pharmacotherapies, and novel research target areas in the treatment of alcohol dependence: a review. Curr Pharm Des. 2011;17(14):1323-32. doi: 10.2174/138161211796150765. PMID 21524263